CLINICAL TRIAL: NCT02886091
Title: Observational Study of Keloids Scars Treated by Shaving and Cryosurgery
Acronym: KELOIDS SCARS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: KELOIDS SCARS
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Keloids Scars
Keywords: Keloids; Shaving; Ears; Cryosurgery; Hypertrophic scars
MeSH Terms: conditions — Keloid; Cicatrix, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Treatment of keloids scars is difficult and controversial. These keloids have a functional and aesthetic impact. A lot of treatment are described with a lot of relapses and aggravation. Authors report outcomes of the treatment with shaving and cryosurgery

ELIGIBILITY:
Inclusion Criteria:

* keloids scars
* treatment of shaving and cryosurgery

Exclusion Criteria:

* immunosuppressive therapy
* chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Keloids scars
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2014-08; Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
size scar | Inclusion and one years after
  reduction size scar

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Trimaille, Study Director — CHRU de Brest
Locations (1):
- CHRU de Brest, Brest, France